CLINICAL TRIAL: NCT04553224
Title: Collection of Clinical and Biometrological Data in Adult Subjects Suffering From Atopic Dermatitis (AD) During a Three-month Period
Brief Title: Collection of Clinical and Instrumental Data in Adult Subjects Suffering From Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POSCORADCOLLECT
Record Dates: First submitted 2020-05-14; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Other): Clinical and instrumental measurements
  Interventions: Other: Clinical evaluations; Other: Non-invasive instrumental measurements; Other: Subject's evaluations

INTERVENTIONS:
Other: Clinical evaluations — SCORAD and target SCORAD
Other: Non-invasive instrumental measurements — TEWL, cutaneous hydration, skin lipidic analysis, colorimetry, hydration index
Other: Subject's evaluations — PO-SCORAD, target PO-SCORAD and subject's questionnaire

SUMMARY:
Atopic dermatitis represents a real challenge in public health as it affects a large percentage of children and adults. Affected individuals must cope with a significant psychosocial burden, in addition to dealing with the medical aspects of the disease.

The purpose of this exploratory study is to collect clinical severity AD data, using PO-SCORAD (self-assessment by the subjects), SCORAD evolution, instrumental measurements and treatment follow up of subjects.

The future objective is to develop a personalised prediction model of AD flares in order to improve management of AD by more accurate severity evaluations by the subject and the physician. Development of a method of early detection of flares will open new treatment pathways for AD management.

DETAILED DESCRIPTION:
This study will be conducted as a French monocentric exploratory study in adults with mild to moderate Atopic Dermatitis, and will be conducted on a maximum 25 included subjects.

The clinical study will include 4 study visits, after inclusion visit, and the maximum duration of the study for each subject will be 3 months : Day 1, Day 29, Day 57, Day 85.

In case of AD flare suspicion, the investigator may recommend a complementary visit. Any complementary visit will be confirmed by investigator according to the subject's information: photographs and PO-SCORAD sent by the subject. If visit is confirmed, it will be scheduled as soon as possible.

The objectives are:

* to collect clinical AD severity data in order to evaluate natural AD evolution with clinical and subject's scales, during a three-month period.
* to collect non-invasive instrumental AD data on a target area and on adjacent area: cutaneous hydration, epidermal barrier conditions and colorimetric parameters on cutaneous erythema
* to examine clinical and instrumental AD data
* to collect illustrative photographs of AD lesions

ELIGIBILITY:
Only most important inclusion and exclusion criteria are listed : those which are study specific.

Inclusion Criteria:

* Subject suffering from Atopic Dermatitis according to the U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis (3).
* Subject with mild to moderate Atopic Dermatitis with 20 <= SCORAD <= 40 at inclusion
* Subject with flare frequency ≥ 4 over the last year
* Subject with a cutaneous target area, allowing the measurements, located on upper or lower limbs and defined as a usual AD flare area according to the subject
* Subject owning a smartphone suitable with the 5.0 downloaded version of PO-Scorad® app
* Subject who agrees to use daily a free mobile app: PO-Scorad®

Exclusion Criteria:

* Subject having received artificial UV exposure or excessive exposure to natural sunlight within the 2 weeks before the inclusion visit or planning to be exposed to excessive or prolonged natural sunlight or UV exposures for the duration of the study
* Subject with a hirsute target area
* Systemic immunosuppressive therapy (excepted systemic corticoids) within 3 months before the inclusion visit or ongoing at inclusion visit.
* Systemic corticoids taken (whatever the number of intake) within 4 weeks before the inclusion visit or ongoing at inclusion visit.
* Phototherapy performed within 4 weeks before the inclusion visit or ongoing at inclusion visit
* Systemic antibiotics taken within 7 days before the inclusion visit or ongoing at inclusion visit.
* Moderate to high-potency topical corticosteroids applied within 7 days on upper or lower limbs before the inclusion visit or ongoing at inclusion visit
* Topical immunomodulators (TIMs), applied within 7 days on upper or lower limbs before the inclusion visit or ongoing at inclusion visit
* Any topical treatment or product applied between the evening before the inclusion visit and the inclusion visit
* Water applied on target area within 4 hours before the inclusion visit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change on clinical evaluation (investigator evaluation) : SCORAD | Day1, Day29, Day57 and Day85
  The SCORAD is a scoring system based on the assessment of extent and intensity in a standardized manner
Change on clinical evaluation (investigator evaluation) : Target SCORAD | Day1, Day29, Day57 and Day85
  Target SCORAD is the sum of all SCORAD objective signs scores: erythema, oedema/papulation, oozing/crusts, excoriation, lichenification and dryness evaluated on a target area
Change on instrumental measurement performed by investigational team : TEWL | Day1, Day29, Day57 and Day85
  TEWL: Transepidermal water loss. TEWL tracks the passage of water through the skin
Change on instrumental measurement performed by investigational team : Lipidic analysis | Day1, Day29, Day57 and Day85
  The proportion of lipids will be analysed on specific bands of infrared spectra by calculation of area under curve of the peaks
Change on instrumental measurement performed by investigational team : cutaneous hydration | Day1, Day29, Day57 and Day85
  Cutaneous hydration evaluated by humidity of the stratum corneum. The measurement is based on capacitance measurement of the stratum corneum.
Change on instrumental measurement performed by investigational team : colorimetric parameter of cutaneous erythema | Day1, Day29, Day57 and Day85
  Evaluation with objective assessment the color of the surface of the skin. Data output will be in the form of the L* a* b* color coordinate system. The a* values (red/ green) will be assessed for quantifying the degree of erythema.
Change on instrumental measurement by subject | each day, during 3 months
  hydration index : mean value measured by a measuring pen on the skin
Change on Subject's evaluations : subject evaluation | each day during 3 months
  PO-SCORAD : a fully validated self-assessment of the AD severity adapted from the SCORAD index; it is available on mobile's phone application.
Change on Subject's evaluation : subject evaluation | on Day1, Day29, Day57 and Day85
  target PO-SCORAD : The target PO-SCORAD is the sum of all PO-SCORAD objective signs scores: dryness of the skin without eczema, redness of the skin affected by eczema, swelling, oozing/ crust, scratching and thickening evaluated on the target area
Change on Subject's evaluation : subject evaluation | once a month
  Subject's questionnaire on lifestyle modifications, as potential flare triggers.

CONTACTS AND LOCATIONS:
Overall Officials: Didier COUSTOU, MD, Principal Investigator
Locations (1):
- Skin Research Centre, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: free mobile app: PO-Scorad® — https://www.poscorad.com/